CLINICAL TRIAL: NCT04339881
Title: NOsocomial Dissemination Risk of SARS-Cov2
Acronym: NODS-Cov2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200417
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, in France, in the context of the SARS Cov2 pandemic,both the number of affected subjects and the number of severe forms requiring hospital care are increasing.

Several nosocomial transmission clusters have already been identified in hospitals (both pediatric and adult) but there is still limited data on the nosocomial spread of SARS-Cov2.

This nosocomial transmission affects both patients and caregivers. It is important to understand the spread of the virus within the hospital. This will help to optimize procedures to prevent transmission to caregivers and hospitalizedpatients not infected with SARS Cov2, and more generally this will contribute to control the spread of SARS Cov2 in the community

DETAILED DESCRIPTION:
It is an observational study without any risk. Every participating service will be investigated for 2 consecutive days .

* At each staff rotation, an individualsensorwill be provided toall thestaff(caregivers, administrative, students etc…) to be worn duringtheirworking hours. Also a sensor will be placed at each patient's bedside.
* In addition, epidemiological data relating to socio-demographic characteristics, profession, protective measures will be collectedfrom hospitalstaff. Also, some data from the 'entrepot des données de santé" regarding individual carepathways in the hospitalwill be extracted.
* A map of the unit, specifying the location of each patient will be made.

ELIGIBILITY:
Inclusion Criteria for patients:

* Informed of the purpose of the study and having expressed his non-opposition or of a relative (if the patient's state of health does not allow it)
* Hospitalized in one of the participating departments

Inclusion criteria for hospital staff:

* Informed of the objective of the study and having expressed his no opposition
* Having daily contact with patients hospitalized in participating departments

Inclusion criteria for patient visitors

* Informed of the purpose of the study and having expressed his non-opposition
* Having daily contacts with patients hospitalized in the participating departments

Exclusion Criteria for evryone (patient, hospital staff and patients visitors) :

* Refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Working caregivers and hospitalized patients in care services dedicated or not to SARS Cov2 (including resuscitation services) in both adult and pediatric hospitals. Investigator will be interested in both adult and child services because the latter present a pauci-symptomatic form so the dynamics of transmission can be different.
Sampling Method: Non-Probability Sample
Enrollment: 2523 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-12 (Actual)

PRIMARY OUTCOMES:
Understanding the dissemination of SARS Cov2 in hospital | 2 days
  In each unit, during 2 days, Patients and all staff (caregivers, administrative, students…) will carry an individualsensorwhich will regularly measure the proximity between 2 sensors

SECONDARY OUTCOMES:
Optimizing hospital strategies to prevent transmission to caregivers and not infected hospitalized patients with SARSCov2 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Didier Guillemot, Garches, France